CLINICAL TRIAL: NCT03208478
Title: A Prospective Comparison of Pain and Quality of Recovery in Patients Undergoing Anterior Cruciate Ligament Reconstruction With Adductor Canal or Femoral Perineural Infusions
Brief Title: Pain Control for Anterior Cruciate Ligament Reconstruction Patients With Adductor Canal or Femoral Perineural Infusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean-Louis Horn, Professor-Med Ctr Line, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 41970
Record Dates: First submitted 2017-06-27; First posted 2017-07-05 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pain, Postoperative; Anterior Cruciate Ligament Injury
MeSH Terms: conditions — Pain, Postoperative; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adductor Canal Nerve Block group (Active Comparator): Adductor Canal perineural catheter placement. Adductor Canal continuous perineural infusion. Ropivacaine 0.2% will be administered at a continuous rate of 5 mL/hour through a perineural catheter placed in the adductor canal. A Nimbus pump (Infutronix) will be delivering the medication.
  Interventions: Procedure: Adductor Canal perineural catheter placement; Device: Nimbus pump (Infutronix)
- Femoral Nerve Block group (Active Comparator): Femoral Nerve perineural catheter placement. Femoral continuous perineural infusion. Ropivacaine 0.2% will be administered at a continuous rate of 5 mL/hour through a perineural catheter placed near the femoral nerve. A Nimbus pump (Infutronix) will be delivering the medication.
  Interventions: Procedure: Femoral Nerve perineural catheter placement; Device: Nimbus pump (Infutronix)

INTERVENTIONS:
Procedure: Adductor Canal perineural catheter placement — Patients will receive an Adductor Canal Block intervention for pain control following ACL reconstructive surgeries.
  Other Names: Adductor Canal block
  Arms: Adductor Canal Nerve Block group
Procedure: Femoral Nerve perineural catheter placement — Patients will have a Femoral perineural catheter placed for pain control following ACL reconstructive surgery.
  Other Names: Femoral Nerve Block
  Arms: Femoral Nerve Block group
Device: Nimbus pump (Infutronix) — This is a FDA approved infusion device that is used in standard of care to store pain medication and to provide patients with continuous pain control medication at a set rate. This pump will be used for both the Adductor Canal and Femoral Nerve block participants.

SUMMARY:
Nerve blocks are used to provide pain control after moderately painful orthopedic surgeries. Anterior Cruciate Ligament (ACL) reconstruction with patellar autograft is a painful orthopedic procedure performed after traumatic injury to the knee. Many patients undergoing ACL reconstruction receive a nerve block as part of their anesthetic care. These blocks can be performed in different locations along the femoral nerve, with advantages and disadvantages to each location. Recently published evidence indicates that there is no short-term difference in pain control between the two commonly-targeted locations ("Adductor Canal" and "Femoral"). However, studies involving patients undergoing total knee arthroplasty indicate that femoral blocks provide better pain control with movement than adductor canal blocks. As many patients undergoing ACL reconstruction use continuous passive motion (CPM) machines as part of rehabilitation starting on post-operative day one, the investigators hypothesize that pain control and quality of recovery in the first 48 hours after surgery will be superior with a continuous femoral block than with a continuous adductor canal block. The investigators plan to study this by randomizing patients presenting for ACL reconstruction to receive either a continuous femoral or continuous adductor canal block (both considered adequate means of pain control), and following them to 48 hours to determine the level of pain, quality of recovery score, opioid use, and CPM compliance.

DETAILED DESCRIPTION:
covery score, opioid use, and CPM compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >18 years
* ASA physical status I, II, or III
* Scheduled for ACL reconstruction surgery with patellar autograft

Exclusion Criteria:

* Pregnancy
* Incarceration
* Age <18
* BMI >35
* Pre-operative opioid use >15 mg morphine equivalents per day
* Inability to communicate with investigators by telephone
* Pre-existing neuropathy of the operative extremity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Pain Score | Post-operative day 2
  Participants will report pain on a numeric rating scale

SECONDARY OUTCOMES:
Quality of Recovery | POD 2
  The Quality of Recovery 15 (QoR 15) is a 15-item questionnaire that is often used to assess how patients are doing in their post-operative course. This survey will be used to assess participants' quality of recovery after ACL reconstructive surgery.
Opioid Use | POD 2
  Total morphine equivalents used through POD 2
CPM compliance | POD 2
  number of hours of reported CPM usage through POD 2

OTHER OUTCOMES:
Quality of Recovery | POD 1
  The Quality of Recovery 15 (QoR 15) is a 15-item questionnaire that is often used to assess how patients are doing in their post-operative course. This survey will be used to assess participants' quality of recovery after ACL reconstructive surgery.
Bolus dose usage | POD 2
  Total volume of patient-administered bolus doses over the course of the infusion
Return to Play | 3 months
  Binary variable, whether patient has returned to normal sports activities
Quadriceps Circumference, percent of baseline | 3 months
  Quadriceps Circumference in cm measured 3 months after surgery, divided by pre-surgery circumference

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis-Horn, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No